CLINICAL TRIAL: NCT03812055
Title: Cellular Pharmacodynamics of Small Molecules in Sanfilippo Disease(s) (MPS3) and Other Lysosomal Storage Disorders
Brief Title: Cellular Pharmacodynamics of Small Molecules in Lysosomal Storage Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 18-LDRTC-02
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lysosomal Storage Diseases
MeSH Terms: conditions — Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LSD: Subjects diagnosed or suspected to have any of the following lysosomal storage diseases: Gaucher disease, Fabry disease, Pompe disease, Mucopolysaccharidoses.
- Control: Subjects with no known lysosomal storage disorder

SUMMARY:
The purpose of this study is to evaluate the effect of small molecule therapy in primary cells derived from patients with lysosomal storage disease. The study will focus on activity of small molecules, in terms of measurements enzymes activity and level of substrates accumulations. Also, the effects of small molecules on cell function, including autophagy-lysosomal pathways, metabolism, mitochondrial function and immune reaction will be investigated.

DETAILED DESCRIPTION:
Lysosomal storage diseases (LSD) often cause severe disability and have a devastating effect on quality of life. The current standard of care of a majority of LSD is enzyme replacement therapy (ERT). ERT, however, becomes less effective during the advanced stages of a disease. Another therapy is substrate reduction therapy (SRT). For example, SRT therapy for Gaucher disease with small molecules acts on ceramide synthesis pathway by decreasing production of the substrate. But, none of the above therapies are effective for treatment of a neuropathic form of LSD. Neurodegenerative changes in the central nervous system are a major problem in Sanfilippo disease. They cause severe disability and behavioral disturbance. This is the main reason for the absence of therapeutic options for MPS3 (Sanfilippo) patients. The future of neuropathic form of LSD therapy may lie in small molecules acting as agents for enzyme-enhancement therapy (EET). EET is based on the ability of small molecules to fold the misfolded mutant enzyme, activate autophagy-lysosomal pathways or mitochondrial function. This treatment approach has the potential to cross the CNS and carries the potential to treat the neurological symptoms of Sanfilippo disease or other types of LSD.

The purpose of this study will evaluate the effect of small molecule therapy in primary cells derived from patients with lysosomal storage disease. The study will be focused on activity of small molecules, in terms of measurements enzymes activity and level of substrates accumulations. Also, the effects of small molecules on cell function, including autophagy-lysosomal pathways, metabolism, mitochondrial function and immune reaction will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Subjects with

1. confirmed diagnosis of any lysosomal storage disorder
2. family members with history of lysosomal storage disorders

Exclusion Criteria:

Subjects excluded from the study include those who:

1. present with severe cognitive deficits impairing decision making
2. are unable to or for whom it is medically unsafe to withdraw from their current medications, such as subjects on SSRI s and other psychoactive drugs. The subjects on SSRIs may be included in the study only with an approval from the prescribing physician to discontinue their medications temporarily for the study.
3. are pregnant or nursing. All women of child bearing potential will undergo a pregnancy test.
4. have a history of neurologic conditions such as stroke or any focal brain lesion that may result in parkinonian manifestations. Individuals with such MRI findings will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed or suspected of having a lysosomal storage disorder and family members of diagnosed patients will be recruited. Informed consent will be obtained prior to the execution of any research procedures.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Effect on enzyme activity | 24 months
  To evaluate the effect of small molecules on level of enzyme activity in primary cells derived from patients using fluorometric enzyme assays.
Effect on substrate accumulation | 24 months
  To evaluate the effect of small molecules on heparin sulfate accumulation and substrate accumulation in primary cells derived from patients using techniques like ELISA and mass spectrometry
Effect on autophagy-lysosomal pathway | 24 months
  To evaluate the effect of small molecules on autophagy-lysosomal functions in primary cells derived from patients using commercially available assays
Effect on mitochondrial functions | 24 months
  To evaluate the effect of small molecules on energy metabolism and mitochondrial functions in primary cells derived from patients using commercially available assay kits
Effect on immune and inflammatory response | 24 months
  Examine the immune and inflammatory response to treatment with small molecules using flow cytometry based immunophenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Margarita M Ivanova, PhD, Principal Investigator — LDRTC; Ozlem Goker-Alpan, MD, Principal Investigator — LDRTC; Renuka Limgala, PhD, Principal Investigator — LDRTC
Locations (1):
- LDRTC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Institute website for more details — http://www.ldrtc.org